CLINICAL TRIAL: NCT06757751
Title: Antidiabetic Potential of Galician High-phenolic Extra Virgin Olive Oils in Patients With Type 2 Diabetes
Brief Title: Antidiabetic Potential of Galician High-phenolic Extra Virgin Olive Oils in Patients With Type 2 Diabetes Mellitus.
Acronym: OILDIABET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacin Biomedica Galicia Sur (Other)
Responsible Party: Principal Investigator, Beatriz Cancho Grande, PhD, Fundacin Biomedica Galicia Sur
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OILDIABET
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): For 24 weeks, subjects in this arm will have their diet supplemented, daily, with an amount of 30 ml of EVOO (Extra Virgin Olive Oil).
  Subjects in this arm will also receive qualitative dietary recommendations for following a healthy diet from the nutritional recommendations for patients with diabetes (Evert et al. (2013). Diabetes Care, 36 (11), 3821-3842.).
  Interventions: Dietary Supplement: EVOO diet supplement
- Control arm (No Intervention): Subjects in this arm will receive qualitative dietary recommendations for following a healthy diet from the nutritional recommendations for patients with diabetes (Evert et al. (2013). Diabetes Care, 36 (11), 3821-3842.).

INTERVENTIONS:
Dietary Supplement: EVOO diet supplement — For 24 weeks, subjects in intervention arm will have their diet supplemented, daily, with an amount of 30 ml of EVOO (Extra Virgin Olive Oil).
  Arms: Intervention arm

SUMMARY:
Since Galician virgin olive oils have a high content of bioactive phenolic compounds and these are attributed to a large part of the healthy properties of the Mediterranean Diet, our starting hypothesis is that these olive oils could attenuate insulin resistance, improving glycemic control in terms of fasting plasma glucose and/or glycated hemoglobin and insulin sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus for at least 1 year prior to inclusion.
* Older than 18 years old
* Current treatment with diet and/or oral hypoglycemic agents (biguanides, thiazolindiones, α-glucosidase inhibitors, iDPP4, aGLP-1, iSGLT2).
* Body mass index ≥ 25 kg/m2 and < 40 kg/ m2.

Exclusion Criteria:

* Patients on treatment with insulin, SU or rapid-acting insulin secretagogues.
* History of severe ketosis or hyperglycemic decompensation.
* Pregnancy, pregnancy planning or breastfeeding.
* Body mass index ≥ 25 kg/m2 and < 40 kg/m2.
* Difficulty or great inconvenience in changing eating habits or a low predicted probability of changing eating habits.
* Serious medical condition that may affect the person's ability to participate in a nutritional intervention study (e.g., digestive disease with fat intolerance, malignant disease, or significant neurological, psychiatric, or endocrine disease).
* Any other medical condition considered to limit survival to less than 1 year.
* Immunodeficiency or HIV positive status.
* Illegal drug use, chronic alcoholism or problematic alcohol use or total daily alcohol intake > 80 g/d.
* Participation in any clinical trial or use of any investigational drug within the past year.
* Patients institutionalized for chronic care.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Glycosylated hemoglobin (HbA1c) | At baseline, at 12 weeks and at 24 weeks
Fasting plasma glucose (FPG) | At baseline, at 12 weeks and at 24 weeks
  mg/dl

SECONDARY OUTCOMES:
Age | Baseline
  Years
Sex at birth | Baseline
  Male/female
Cardiovascular Risk Factors | Baseline
  Cardiovascular risk factors from the following list will be indicated:
  Arterial hypertension: Yes/No Dyslipidemia: Yes/No
  Smoking:
  Non-smoker Current smoker Recent ex-smoker (<1year) Former smoker (≥1year)
Hepatic dysfunction | Baseline
  Yes/No
Previous heart disease | Baseline
  Yes/No
Heart failure | Baseline
  Yes/No
Coronary Heart Disease | Baseline
  Yes/No
  If yes, answer the following questions:
  * Acute coronary syndrome: Yes/No
  * Coronary revascularization: Yes/No
Concomitant pharmacological treatment | Baseline
  The concomitant pharmacological treatment will be indicated by marking the appropriate one in the following list:
  Diuretics: Yes/No Mineralcorticoid receptor antagonists: Yes/No ACE inhibitors: Yes/No ARBs2: Yes/No Sacubitril/Valsartan: Yes/No Ivabradin: Yes/No Statins: Yes/No AntiPCSK9: Yes/No Ezetimibe: Yes/No Fibrates: Yes/No Antiaggregants: Yes/No Anticoagulants: Yes/No Beta-blockers: Yes/No Calcium antagonists: Yes/No Antiarrhythmics: Yes/No
Antidiabetic treatment | Baseline
  Antidiabetic treatment: Yes/No
  If Yes, will indicate which of the following list:
  Metformin: Yes/No Sulfonylurea: Yes/No I-DPP4: Yes/No I-SGLT2: Yes/No ArGLP1: Yes/No Pioglitazone: Yes/No Insulin: Yes/No
  If insulin is "Yes", which type of dose from the following list will be indicated:
  Basal (1); Two-dose NPH or premixes (2); Basal-bolus (3); Total daily dose: IU/day
Systolic Blood Pressure | At baseline, at 12 weeks and at 24 weeks
  mm Hg
Diastolic blood pressure | At baseline, at 12 weeks and at 24 weeks
  mm Hg
Heart rate | At baseline, at 12 weeks and at 24 weeks
  beats/minute
Weight | At baseline, at 12 weeks and at 24 weeks
  kg
Heigth | Baseline
  cm
Body Mass Index (BMI) | Baseline
  kg/m2
Urinary albumin excretion (UAE) | At baseline, at 12 weeks and at 24 weeks
  mg/24 h
Estimated Average Plasma Glucose | At baseline, at 12 weeks and at 24 weeks
  mg/dl
Fasting Insulin | At baseline, at 12 weeks and at 24 weeks
  µU/ml
Homeostatic Model Assessment for beta-cell function (HOMA-B) | At baseline, at 12 weeks and at 24 weeks
Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) | At baseline, at 12 weeks and at 24 weeks
  Adimensional
N-terminal pro-B-type natriuretic peptide (NT-proBNP) | At baseline, at 12 weeks and at 24 weeks
  pg/ml
Total cholesterol | At baseline, at 12 weeks and at 24 weeks
  mg/dl
LDL-C HDL-C, mmol/l | At baseline, at 12 weeks and at 24 weeks
  mg/dl
HDL-C | At baseline, at 12 weeks and at 24 weeks
  mg/dl
Triglycerides (TG) | At baseline, at 12 weeks and at 24 weeks
  mg/dl
Dietetic education | At baseline, at 12 weeks and at 24 weeks
  Visit with Dietitian: Yes/No
Cardiovascular events | At 12 weeks and at 24 weeks
  It will be indicated if cardiovascular events have occurred: Yes/No

CONTACTS AND LOCATIONS:
Locations (1):
- Beatriz Cancho Grande, Ourense, Spain